CLINICAL TRIAL: NCT02459093
Title: Comparison of Subcuticular Suture Type in Post-Cesarean Wound Complications
Brief Title: Subcuticular Suture for Cesarean Skin Incision Closure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, David Garry, Maternal Fetal Medicine Specialist, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-4655
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Complications; Cesarean Section; Surgical Wound Infection
Keywords: wound complications
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- poliglecaprone 25 suture (Experimental): Subcuticular skin approximation with poliglecaprone 25 suture at cesarean birth surgery
  Interventions: Device: poliglecaprone 25 suture
- polyglactin 910 suture (Experimental): Subcuticular skin approximation with polyglactin 910 suture at cesarean birth surgery
  Interventions: Device: polyglactin 910 suture

INTERVENTIONS:
Device: poliglecaprone 25 suture — cesarean delivery incision closure with poliglecaprone 25 suture
  Other Names: MONOCRYL Suture (poliglecaprone 25 suture)
  Arms: poliglecaprone 25 suture
Device: polyglactin 910 suture — cesarean delivery incision closure with polyglactin 910 suture
  Other Names: VICRYL Suture (polyglactin 910 suture)
  Arms: polyglactin 910 suture

SUMMARY:
A comparison of the type of suture used for cesarean skin incision approximation and the subsequent rate of wound complications has not been widely studied. Investigators seek to compare poliglecaprone 25 and polyglactin 910 suture used in a subcuticular skin closure in Pfannenstiel incisions during cesarean birth and determine the subsequent wound complication rates (SSI, hematoma, seroma, wound separation).

DETAILED DESCRIPTION:
In the United States cesarean delivery rates in 2012 were 32.8%. The incidence of wound complications post-cesarean delivery has been quoted to be anywhere from 3-30%. Wound complications can include surgical site infection (SSI), hematoma, seroma, and wound separation. Risk factors for wound complications include elevated body mass index (BMI), prolonged duration of surgery, maternal diabetes, coexisting infection (chorioamnionitis), anemia, and increasing number of prior cesarean deliveries. The majority of cesarean deliveries are performed through a suprapubic low-transverse skin incision (Pfannenstiel incision). The incidence of wound complication post-cesarean comparing suture and staple skin closure has been extensively studied with the over all conclusion recommending suture skin closer.

A comparison of the type of suture used for skin closer and wound complication has not been widely studied. Vats et al. compared three types of suture material in post-cesarean wound complication and found statistical difference in wound discomfort, swelling and induration, wound discharge, and wound dehiscence. Their quoted wound complication rate was as high as thirty-three percent. Although, their study population was limited to emergent cesarean deliveries, the sample size was small, and their method of randomization was not explained.

Physiologic wound healing involves five steps: inflammation, granulation, epithelialization, wound contraction, and scar maturation. These biologic processes overlap in occurrence but happen in a defined order. Investigators hypothesize that suture materials with differing profiles will have different effects on these biologic processes. The two most widely used sutures for low-transverse cesarean skin incision closure in our institution are poliglecaprone 25 and polyglactin 910. Poliglecaprone 25 (monocryl) is a monofilament suture with an absorption profile of 91-119 days. Polyglactin 910 (coated vicryl) is a braided suture with an absorption profile of 56-70 days. Given the difference in profile for each suture and the physiologic wound healing process investigators question which would be more effective for wound healing.

The purpose of the study:

1. To compare poliglecaprone 25 and polyglactin 910 suture in Pfannenstiel incision closure for prevention of wound complication (SSI, hematoma, seroma, wound separation).
2. To determine if risk factors for wound complication should guide the choice of suture used for closure of Pfannenstiel incision.

Methods Patient enrollment will occur during their admission to labor and delivery. Patients will be approached if they meet the enrollment criteria. If they agree to participate in the trial a pre-randomized sequentially numbered, opaque, sealed envelope will be assigned to them and opened at the time of cesarean delivery which will assign the surgical suture to be used for skin closure.

Inclusion criteria for the trial:

1. Gestational age of 37 completed weeks or greater based on their estimated due date calculated from last menstrual period or early ultrasound.
2. Scheduled cesarean delivery or...
3. Non-emergent cesarean delivery

Patients participating will be undergoing either:

1. Scheduled cesarean delivery
2. Non-emergent cesarean delivery

Non-emergent cesarean delivery will be defined as an indicated cesarean delivery based on obstetrical criteria without significant fetal heart tracing abnormalities. This would include women diagnosed with a labor dystocia or arrest of labor, failed labor induction, fetal malpresentation in labor (i.e. breech presentation) or any other non-emergent indication for cesarean delivery in which there is no immediate danger to mother or fetus.

The following exclusion criteria will be used:

1. Urogenital tract infection within 2 weeks prior to surgery
2. Chronic oral or injectable steroid use (> 2 weeks)
3. Emergency cesarean delivery (need to deliver immediately due to a maternal or fetal indication)
4. Vertical skin incision
5. Participation in another research study

The patients will be randomized after informed consent is obtained into two groups.

Group 1: Incision closure with poliglecaprone 25 suture Group 2: Incision closure with polyglactin 910 suture

Randomization for the study will be generated using www.randomization.com, in blocks of 6 and 10 prior to the start of enrollment for the trial. Sequentially numbered, opaque, sealed envelopes will contain the surgical suture to be used for skin closure, poliglecaprone 25 or polyglactin 910.

Surgical preparation will follow departmental protocol. Once the patient is randomized to a suture group the corresponding suture will be pulled and placed on the sterile field for use after completion of the cesarean in accordance to manufacturer's guidelines. Cesarean delivery will occur following the technique of the surgeon. Maternal demographics to be obtained will include BMI, gestational age, pre and postoperative day #1 complete blood count, estimated blood loss, type of preoperative skin preparation, surgical time from skin incision to closure, birth weight, Apgar scores, newborn outcome, indication for cesarean delivery, medical history and any antenatal complications, past surgical history, postoperative course, and intraoperative or postoperative complications. Wound complication will be defined as wound separation of ≥ 1 cm in length, hematoma or seroma (serous fluid collection or subcutaneous blood collection), and surgical site infection defined by the Center for Disease Control (CDC) guidelines. The primary outcome will include a composite finding of a wound complication in the 30 day period post-operatively.

All patients will be followed until the routine postpartum visit occurs at 6-8 weeks following delivery with their primary prenatal care provider. Postpartum visit information will be extracted from the medical record. All patients will receive a follow up telephone call at post-operative day 30 or greater to monitor any post-operative complications as listed above.

An alert notification will be placed in each patient's medical record that they are enrolled in this study and close monitoring and documentation of the cesarean incision is necessary. The definition of wound complication as listed in the first paragraph above will be included in the alert notification to standardize reporting for each patient.

Recruitment Mechanisms Clinicians will ask patients during admission to labor and delivery after they meet enrollment criteria whether they are interested in the study. Consent will then be obtained by the research clinicians.

Informed Consent Patient consent will occur on admission to the labor and delivery unit. The capacity of each patient to provide ethically adequate informed consent will be assessed by the PI or his designee. It is possible that patients will be enrolled during labor prior to cesarean section if not in significant pain although the majority of patients will be presenting for scheduled cesarean sections prior to labor. Consent will be obtained from women in active labor after labor analgesia has occurred. Emergency cesareans are excluded.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 37 completed weeks or greater based on their estimated due date calculated from last menstrual period or early ultrasound.
* Patients participating will be undergoing either:

  * Scheduled cesarean delivery
  * Non-emergent cesarean delivery

Exclusion Criteria:

* Urogenital tract infection within 2 weeks prior to surgery
* Chronic oral or injectable steroid use (> 2 weeks)
* Emergency cesarean delivery (need to deliver immediately due to a maternal or fetal indication)
* Vertical skin incision
* Active participation in another research study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Garry, DO, Principal Investigator — Montefiore Medical Center / Einstein College of Medicine
Locations (2):
- United States (2):
  - Montefiore Medical Center Weiler Division, The Bronx, New York
  - Montefiore Medical Center Wakefield Division, The Bronx, New York

REFERENCES:
- [Background] Vats U, Pandit Suchitra N. Comparison of Efficacy of Three Suture Materials, i.e., Poliglecaprone 25, Polyglactin 910, Polyamide, as Subcuticular Skin Stitches in Post-Cesarean Women: A Randomized Clinical Trial. J Obstet Gynaecol India. 2014 Feb;64(1):14-8. doi: 10.1007/s13224-013-0448-5. Epub 2013 Sep 4. PMID 24587600
- [Background] Nuthalapaty FS, Lee CM, Lee JH, Kuper SG, Higdon HL 3rd. A randomized controlled trial of early versus delayed skin staple removal following caesarean section in the obese patient. J Obstet Gynaecol Can. 2013 May;35(5):426-433. doi: 10.1016/S1701-2163(15)30933-6. PMID 23756273
- [Background] Mourad M, Silverstein M, Bender S, Melka S, Klauser CK, Gupta S, Saltzman DH, Rebarber A, Fox NS. The effect of maternal obesity on outcomes in patients undergoing tertiary or higher cesarean delivery. J Matern Fetal Neonatal Med. 2015 Jun;28(9):989-93. doi: 10.3109/14767058.2014.941284. Epub 2014 Jul 24. PMID 25058127
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Mackeen AD, Khalifeh A, Fleisher J, Vogell A, Han C, Sendecki J, Pettker C, Leiby BE, Baxter JK, Sfakianaki A, Berghella V. Suture compared with staple skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1169-1175. doi: 10.1097/AOG.0000000000000227. PMID 24807325
- [Background] Corbacioglu Esmer A, Goksedef PC, Akca A, Akbayir O, Dagdeviren H, Turan GY, Yarsilikal F. Role of subcutaneous closure in preventing wound complications after cesarean delivery with Pfannenstiel incision: a randomized clinical trial. J Obstet Gynaecol Res. 2014 Mar;40(3):728-35. doi: 10.1111/jog.12229. PMID 24738117
- [Background] Martin JA, Hamilton BE, Osterman MJ, Curtin SC, Matthews TJ. Births: final data for 2012. Natl Vital Stat Rep. 2013 Dec 30;62(9):1-68. PMID 25671704
- [Result] Buresch AM, Van Arsdale A, Ferzli M, Sahasrabudhe N, Sun M, Bernstein J, Bernstein PS, Ngai IM, Garry DJ. Comparison of Subcuticular Suture Type for Skin Closure After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Sep;130(3):521-526. doi: 10.1097/AOG.0000000000002200. PMID 28796687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Poliglecaprone 25 Suture | Polyglactin 910 Suture
Started | 275 | 275
Completed (Received treatment and completed 30 day follow-up) | 263 | 257
Not Completed | 12 | 18
Not completed — Protocol Violation | 6 | 11
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Poliglecaprone 25 Suture | Polyglactin 910 Suture | Total
Number analyzed (Participants) | 263 | 257 | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.4) | 31.2 (5.4) | 31.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 257 | 520
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 17 | 35
  African American | 64 | 61 | 125
  Hispanic | 128 | 130 | 258
  Asian | 17 | 11 | 28
  Other | 14 | 26 | 40
  Missing | 22 | 12 | 34
Cesarean delivery with labor [Count of Participants; unit: Participants]
  Scheduled or no labor | 224 | 207 | 431
  Any labor | 39 | 50 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complications (Surgical Site Infection (SSI), Hematoma, Separation, Seroma, Etc)
Description: Any wound disruption, fluid accumulation, separation, all CDC defined stages of surgical site infection (SSI)
Time Frame: 30 days
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Poliglecaprone 25 Suture | Polyglactin 910 Suture
Number analyzed (Participants) | 263 | 257
Participants
  Composite wound | 23 | 37
  Surgical Site Infection | 16 | 25
  Hematoma | 1 | 3
  Seroma | 2 | 1
  Separation | 7 | 13
Statistical Analysis 1: Comparison: Poliglecaprone 25 Suture vs Polyglactin 910 Suture; Test type: Superiority; p = 0.04, Chi-squared; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.37 to 0.99]

2. Primary Outcome: Number of Participants With Wound Complications (Surgical Site Infection (SSI), Hematoma, Separation, Seroma, Etc)
Description: Any wound disruption, fluid accumulation, separation, all CDC defined stages of surgical site infection (SSI)
Time Frame: 30 days
Population: As treated
Measure: Count of Participants; unit: Participants
Arm/Group | Poliglecaprone 25 Suture | Polyglactin 910 Suture
Number analyzed (Participants) | 265 | 217
Participants
  Composite wound | 22 | 30
  Surgical Site Infection | 16 | 20
  Hematoma | 1 | 2
  Seroma | 1 | 2
  Separation | 8 | 8
Statistical Analysis 1: Comparison: Poliglecaprone 25 Suture vs Polyglactin 910 Suture; Test type: Superiority; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.60, 95% CI 2-sided [0.36 to 1.01]

ADVERSE EVENTS:
Arm/Group | Poliglecaprone 25 Suture | Polyglactin 910 Suture
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/257
Serious Adverse Events (participants affected / at risk) | 0/263 | 0/257
Other Adverse Events (participants affected / at risk) | 0/263 | 0/257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No